CLINICAL TRIAL: NCT01007188
Title: Energy Value of Macronutrients From Almonds and Mechanisms of Nutrient Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Collaborators: Almond Board of California (Other)
Responsible Party: David J. Baer, Ph. D., Research Leader, Food Components and Health Laboratory, USDA-ARS, BHNRC
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2009-412
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: almond; nuts; energy value; cardiovascular disease; phytonutrient; gene expression; energy value of almonds; energy
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Alkalies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1.5PD (Active Comparator): average American diet plus 1.5 oz per day almonds
  Interventions: Other: 1.5PD almonds
- Base (Other): average American diet without almonds
  Interventions: Other: Base (without almonds)
- 3.0PD (Active Comparator): average American diet plus 3.0 oz per day almonds
  Interventions: Other: 3.0PD almonds

INTERVENTIONS:
Other: 1.5PD almonds — average American diet plus 1.5 oz per day almonds
  Arms: 1.5PD
Other: 3.0PD almonds — average American diet plus 3.0 oz per day almonds
  Arms: 3.0PD
Other: Base (without almonds) — average American diet without almonds
  Arms: Base

SUMMARY:
The U.S. Department of Agriculture (USDA) wants to learn more about the number of calories in almonds and the mechanisms of the health effects of almonds. Epidemiologic studies have demonstrated an inverse or no relationship between nut consumption and body weight, despite the fact that nuts are an energy dense food. Intervention studies have shown that consumption of nuts has no effect on body weight or an effect that is significantly less than predicted. Fecal analyses in studies with peanuts, almonds, and pecans have found increased fecal fat and energy loss with nut consumption; however studies with almonds are lacking.

DETAILED DESCRIPTION:
The objective of this study is to measure the energy value of almonds in the human diet and study molecular mechanisms that may help explain the beneficial health effects of almonds.

Epidemiologic studies have demonstrated an inverse or no relationship between nut consumption and body weight, despite the fact that nuts are an energy dense food. Intervention studies have shown that consumption of nuts has no effect on body weight or an effect that is significantly less than predicted. Fecal analyses in studies with peanuts, almonds, and pecans have found increased fecal fat and energy loss with nut consumption; however studies with almonds are lacking.

Previous studies have suggested that nut consumption imparts a variety of health benefits, including reduction of cardiovascular disease and improved satiety. However, studies of almonds are extremely limited. The aim of this study is to determine the energy value of almonds in the human diet and to probe mechanisms by which almonds impart health benefits. The metabolizable energy value of almond nuts will be calculated based on the chemical composition and energy content of the consumed diet and excreta. This will provide a better estimate of the energy value of almonds than simply calculating energy value based on Atwater factors. In addition to determining the energy value of almonds, we will evaluate the effects of almond-rich diets on plasma phytonutrient levels and on gene expression changes to determine what protective mechanisms are activated by almond consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 65 years at beginning of study
* BMI between 20 and 38 kg/m2
* Fasting glucose < 126 mg/dl
* Blood pressure < 160/100 (controlled with certain medications)
* Fasting total blood cholesterol < 280 mg/dl
* Fasting triglycerides < 300 mg/dl

Exclusion Criteria:

* Presence of kidney disease, liver disease, gout, hyperthyroidism, untreated or unstable hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* History of bariatric or certain other surgeries related to weight control
* Smokers or other tobacco users (during 6 months prior to the start of the study)
* Antibiotic use during the intervention or for 3 weeks prior to any intervention period
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Volunteers who have lost 10% of body weight within the last 12 months or who plan to initiate a weight loss program during the next 10 months
* Known (self-reported) allergy or adverse reaction to pistachios or other nuts
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
to measure the energy value of almonds in the human diet | 3 weeks

SECONDARY OUTCOMES:
to study molecular mechanisms that may help explain the beneficial health effects of almonds | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David J Baer, Ph. D., Principal Investigator — USDA Beltsville Human Nutrition Research Center
Locations (1):
- USDA-ARS, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

REFERENCES:
- [Derived] Novotny JA, Gebauer SK, Baer DJ. Discrepancy between the Atwater factor predicted and empirically measured energy values of almonds in human diets. Am J Clin Nutr. 2012 Aug;96(2):296-301. doi: 10.3945/ajcn.112.035782. Epub 2012 Jul 3. PMID 22760558